CLINICAL TRIAL: NCT01756664
Title: The Use of Sunscreen Starting on the First Day After Ablative Fractional Skin Resurfacing - A Pilot Study.
Brief Title: The Use of Sunscreen Starting on the First Day After Ablative Fractional Skin Resurfacing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Siriraj-Eucerin01; SI402/2012 (Other: Faculty of Medicine Siriraj Hospital, Mahidol University)
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-08

CONDITIONS: PIH
MeSH Terms: interventions — Sunscreening Agents; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Vaseline has been used on the first day after laser treatment
  Interventions: Other: Vaseline
- Sunscreen (Active Comparator): Sunscreen has been used on the first day after laser treatment
  Interventions: Other: Sunscreen

INTERVENTIONS:
Other: Sunscreen
  Arms: Sunscreen
Other: Vaseline
  Arms: Control

SUMMARY:
- The use of sunscreen on the first day after fractional ablative skin resurfacing may reduce the risk of post-inflammatory hyperpigmentation

DETAILED DESCRIPTION:
* The use of sunscreen on the first day after fractional ablative skin resurfacing may reduce the risk of post-inflammatory hyperpigmentation (PIH)
* Therefore, we conducted the study to evaluate the efficacy of the use of sunscreen on the first day after fractional ablative skin resurfacing in reducing the risk of PIH.

ELIGIBILITY:
Inclusion Criteria:

* Patients who want to receive fractional ablative laser resurfacing for acne scars

Exclusion Criteria:

* Pregnancy
* Lactation
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Melanin Index | 3 Month

SECONDARY OUTCOMES:
Erythema Index | 3 Months

OTHER OUTCOMES:
Transepidermal Water Loss | 1 Week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand